CLINICAL TRIAL: NCT01365364
Title: Dopamine Transporter Density Profiles Assessed by Tc-TRODAT and SPECT in Patients With Periodic Limb Movements
Brief Title: Dopamine Transporter Density Profiles in Patients With Periodic Limb Movements
Acronym: DOPATRANSPLM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Marco Tulio de Mello, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CEP0546/08
Record Dates: First submitted 2011-05-16; First posted 2011-06-03 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2011-05

CONDITIONS: Periodic Limb Movements in Sleep
Keywords: PLM; dopamine; physical exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PLM group (Active Comparator): Individuals with increased periodic leg movement index (>5)
  Interventions: Behavioral: Aerobic Physical Exercise
- Non-PLM group (Active Comparator): Individuals with PLM index <5
  Interventions: Behavioral: Aerobic Physical Exercise

INTERVENTIONS:
Behavioral: Aerobic Physical Exercise — All individuals were submitted to physical exercise reaching maximum effort
  Other Names: Acute Physical Exercise: Maximal Exercise Test
  Arms: PLM group
Behavioral: Aerobic Physical Exercise — All individuals were submitted to physical exercise reaching maximum effort
  Other Names: Acute Physical Exercise: Maximal Exercise Test

SUMMARY:
Restless legs syndrome and periodic limb movement (PLM)are sleep-related movement disorders and studies have shown changes in striatal dopaminergic activity in patients with these disorders. Physical exercise has been shown to improve the symptoms of restless legs syndrome and PLM, as has treatment with dopamine agonists. However, the mechanism by which physical exercise acts as a non-pharmacological treatment in improving symptoms of restless legs syndrome and PLM remains unknown. The investigators evaluated dopamine transporter density profiles in 16 sedentary patients (control and experimental - with PLM, groups) and the influence of acute physical exercise on its concentration after a maximal exercise test. Each patient underwent baseline polysomnography to evaluate sleep patterns and PLM index values. After obtaining the polysomnography baseline, the single photon emission computer tomography baseline was determined. Subsequently, the volunteers performed a maximal exercise test in the morning, followed by a single photon emission computer tomography two hours later and polysomnography that night, to assess the effect of acute physical exercise on dopamine transporter and sleep patterns. The results showed significant lower dopamine transporter baseline densities in the striatum region for the experimental group. The results also showed a significant reduction in the periodic leg movement rate in the experimental group and a significant increased percentage of stage-1 non-REM sleep in both groups after maximal exercise test. Significant differences between the groups were only observed for Stage 2 sleep and slow wave sleep. Our results show that patients with PLM had a lower dopamine transporter density in the left putamen region compared to the control group and an acute physical exercise (maximal exercise test) did not alter this profile, providing evidence that this improvement is the result of chronic physical exercise.

DETAILED DESCRIPTION:
Experimental Design Each volunteer (in both control and experimental groups) underwent Polysomnography (PSG) adaptation. After one week, a baseline cerebral SPECT was performed (1-3pm) and a baseline PSG was performed that night to evaluate the sleep pattern and the PLM index. Subsequently (after one week), each subject underwent a maximal exercise test (MET) in the morning (11am to 1pm) after which SPECT examination was performed in the afternoon (1-3 pm). A PSG was then performed that night to evaluate the effect of acute exercise on DAT density and sleep pattern (Figure 1).

ELIGIBILITY:
Inclusion Criteria:

* With and without PLM,
* no other health problems,
* sedentary

Exclusion Criteria:

* Other clinical and neurological conditions,
* continuous pharmacological treatment

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Dopamine Transporter Density Measurement | Baseline and after 5 hours of exercise effort measurements
  Dopamine Transporter Density Measurement assessed by SPECT using TRODAT-1

SECONDARY OUTCOMES:
Exercise Effort Maximum | 1 week after baseline SPECT
  Exercise Effort VO2 maximum measurement

CONTACTS AND LOCATIONS:
Overall Officials: Marco Tulio Mello, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Centro de Estudos em Psicobiologia e Exercicio, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Earley CJ, Kuwabara H, Wong DF, Gamaldo C, Salas R, Brasic J, Ravert HT, Dannals RF, Allen RP. The dopamine transporter is decreased in the striatum of subjects with restless legs syndrome. Sleep. 2011 Mar 1;34(3):341-7. doi: 10.1093/sleep/34.3.341. PMID 21358851
- [Result] Mrowka M, Jobges M, Berding G, Schimke N, Shing M, Odin P. Computerized movement analysis and beta-CIT-SPECT in patients with restless legs syndrome. J Neural Transm (Vienna). 2005 May;112(5):693-701. doi: 10.1007/s00702-004-0217-9. Epub 2004 Oct 27. PMID 15517434
- [Result] Wetter TC, Eisensehr I, Trenkwalder C. Functional neuroimaging studies in restless legs syndrome. Sleep Med. 2004 Jul;5(4):401-6. doi: 10.1016/j.sleep.2004.01.009. PMID 15223000